CLINICAL TRIAL: NCT04624906
Title: A Multi-Center, Open-Label, Single-Arm Phase II Trial of Bendamustine, Rituximab and the Second Generation BTK Inhibitor Acalabrutinib in Previously Untreated Waldenstrom's Macroglobulinemia
Brief Title: Bendamustine, Rituximab and Acalabrutinib in Waldenstrom's Macroglobulinemia
Acronym: BRAWM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3242
Record Dates: First submitted 2020-10-23; First posted 2020-11-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Waldenstrom Macroglobulinemia; WM; Acalabrutinib; Waldenstrom; Macroglobulinemia; BTK inhibitor; BTK; Bruton's Tyrosine Kinase; First line treatment; BRAWM
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — acalabrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Intervention Model Description: Bendamustine, Rituximab and Acalabrutinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm intervention (Experimental): 100 mg Acalabrutinib (ACP-196) oral capsules twice daily for 1 year
  Bendamustine and rituximab will be given for 6 x 28-day cycles. Bendamustine will be given intravenously at 90 mg/m2 on days 1 and 2 of each cycle. Rituximab will be given on day 1 of each cycle (375 mg/m2 intravenously for the first cycle and 1400 mg subcutaneously OR 375 mg/m2 intravenously for subsequent cycles (as per institutional procedures).
  Interventions: Drug: Acalabrutinib; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — 100 mg oral capsules twice daily for 1 year
  Other Names: Calquence
Drug: Bendamustine — 90 mg/m2 on days 1 and 2 of each cycle.
  Other Names: Treanda
Drug: Rituximab — day 1 of each cycle (375 mg/m2 intravenously for the first cycle and 1400 mg subcutaneously OR 375 mg/m2 intravenously for subsequent cycles (as per institutional procedures).
  Other Names: Rituxan

SUMMARY:
This is a multi-centre, open label, single-arm, phase II clinical trial in untreated patients with Waldenstrom's Macroglobulinemia. Symptomatic, previously untreated patients will receive SOC bendamustine and rituximab for 6 28-day cycles. Bendamustine will be given intravenously at 90 mg/m2 on days 1 and 2 of each cycle. Rituximab will be given on day 1 of each cycle (375 mg/m2 intravenously for the first cycle and 1400 mg subcutaneously OR 375 mg/m2 intravenously for subsequent cycles (as per institutional procedures)). Concomitantly, participants will receive 100 mg of the investigational product, Acalabrutinib, orally for 1 year (365 days) at 100 mg BID.

DETAILED DESCRIPTION:
This is a multi-centre, open label, single-arm, phase II clinical trial in untreated patients with WM. Patients will require a biopsy to confirm the pathology and molecular testing for MYD88, CXCR4 and P53 mutations. A bone marrow aspiration and biopsy will be performed to document WM and MRD. Participants will be classified into clinical risk categories based on the International Prognostic Scoring (IPS) System for WM. Symptomatic, previously untreated patients will receive SOC bendamustine and rituximab for 6 28-day cycles. Bendamustine will be given intravenously at 90 mg/m2 on days 1 and 2 of each cycle. Rituximab will be given on day 1 of each cycle (375 mg/m2 intravenously for the first cycle and 1400 mg subcutaneously OR 375 mg/m2 intravenously for subsequent cycles (as per institutional procedures)).

Concomitantly, participants will receive 100 mg of the investigational product, Acalabrutinib, orally for 1 year (365 days) at 100 mg BID. Patients will have pre-treatment computed tomography (CT) scans, and CT scans at 7, 12 and 18 months. Best objective response will be documented using the criteria from the Sixth International Workshop on Waldenstrom's Macroglobulinemia. Assessment of metabolic uptake by positron emission tomography (PET) scan is not considered appropriate for WM as WM usually do not take up fluorodeoxyglucose (FDG). Patients with WM will also have disease assessed using measurements of serum IgM, serum protein electrophoresis (SPE), immunofixation (IFA), and viscosity assessments measured serially. A bone marrow aspiration and biopsy will be done before treatment and at response assessment at cycle 6 and will be repeated if positive. Durability of response will also be assessed at 18 months.

Participants will be followed by extended follow-up by telephone for up to 6 years to obtain data on the secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Have biopsy proven Waldenstrom's macroglobulinemia, (biopsy from within 3 months (+/- 7 days) prior to Day 1).
2. Have not received any systemic treatment for the disease (plasmapheresis, involved field radiation or corticosteroids (for contrast enhanced studies and to acutely control disease-related symptoms or as chemotherapy premedication)) are allowed.
3. Be willing and able to provide written informed consent for the trial.
4. Male or female >=18 years of age on day of signing informed consent and of any racial or ethnic group.
5. Have at least one measurable site of disease based on Cheson Criteria (Appendix C) using standard CT imaging or a quantifiable IgM paraprotein that is two times the upper limit of normal.
6. Have symptomatic or impending symptomatic disease or evidence of hematologic or biochemical compromise related to the lymphoma.
7. Have a performance status of 0-2 on the ECOG Performance Scale.
8. Demonstrate adequate organ function as defined in Table 2. Adequate organ function must be confirmed within 72 hours prior to start of treatment. Patients with abnormal liver enzymes of up to 5 times the upper limit of normal and/or reduced glomerular filtration rate (GFR) or estimated glomerular filtration rate (eGRF) of ≥ 30 mL/min/1.73 m2can be considered for enrolment.
9. A life expectancy > 6 months in the opinion of the investigator.
10. Female subject of childbearing potential should have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication (day 1).
11. Female subjects of childbearing potential should be willing to use 2 highly effective methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study until 2 days post-last dose of acalabrutinib, 4 weeks post-last dose of bendamustine, and 12 months post-last dose of rituximab. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
12. Male subjects should agree to use a highly-effective method of contraception starting with the first dose of study therapy until 2 days post-last dose of acalabrutinib, 6 months post-last dose of bendamustine, and 12 months post-last dose of rituximab.
13. Ability to comply with protocol requirements.

Exclusion Criteria:

1. Previous systemic therapy for WM (other than described in the inclusion criteria).
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 21 days of the first dose of treatment (SD1).
3. Patient is being planned for consolidative autologous stem cell transplant (ASCT).
4. Is on warfarin anti-coagulation
5. Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids 7 days prior to the start of treatment are eligible.

5. Has clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac diseases as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 480 msec at screening. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.

6. Has clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac diseases as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 480 msec at screening. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.

7. Has hypertension that cannot be controlled with anti-hypertensives. 8. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 35 days prior to the first dose of trial treatment (SD1), except that used as pre-medication for chemotherapy or contrast-enhanced studies are eligible. Subjects may be on physiologic doses of replacement prednisone or equivalent doses of corticosteroid (<10 mg daily).

9. Has a known history of active TB (Bacillus Tuberculosis). 10. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.

11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for their CNS disease for at least 35 days prior to trial treatment.

12. Has history of active autoimmune disease that has required systemic immune suppressive treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.

13. Has known history of, or any evidence of active, non-infectious pneumonitis that has required treatment in the last five years.

14. Has an active infection requiring systemic therapy. Note: Subjects completing a course of antibiotic for acute infection 7 days prior to SD1 and who do not experience a recurrence of symptoms or fever are eligible.

15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

17. Is breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with screening visit to 2 days post last dose of acalabrutinib, 4 weeks post last dose of bendamustine and 12 months post last dose of rituximab.

18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).

19. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., Hepatitis C Virus (HCV) RNA [qualitative] is detected). Evidence of Hepatitis B surface antigen or Hepatitis B DNA are exclusion criteria. Participants with positive hepatitis B core antibody (HBcAb) can be enrolled only if confirmatory negative Hepatitis B Virus (HBV) DNA levels is obtained by polymerase chain reaction (PCR) AND the patient is on Hepatitis B prophylaxis before the first dose of study drug.

20. Serious intercurrent chronic or acute illness, such as hepatic disease, or other illness considered by the investigator as an unwarranted high risk for an investigational product.

21. History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.

22. History of bleeding diathesis (e.g., hemophilia, von Willebrand disease). 23. Requires treatment with a strong* cytochrome P450 3A (CYP3A) inhibitor or within 1 week or a strong CYP3A inducer within 3 weeks of the first dose of study drug is prohibited. *boceprevir, clarithromycin, conivaptin, indinavir, itraconazole, ketoconazole, lopin/ritonavir combination, fluconazole, izavuconazole, mibefradil, nefazodone, nelfinavir, saquinavir, posaconazole, ritonavir, telaprevir, telithromycin, voriconazole, carbamazepine, phenytoin, rifampin or St. John's wort.

24. Received a live virus vaccination within 28 days of first dose of study drug.

25. Major surgical procedure within 30 days before the first dose of study drug. Note: if a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.

26. Refractory nausea and vomiting, inability to swallow the formulated product, or malabsorption syndrome; chronic gastrointestinal disease, gastric restrictions, or bariatric surgery such as gastric bypass partial or complete bowel obstruction, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Best combined complete response (CR) and very good partial response (VGPR) | through study completion, an average of 1 year - cycle 7, 12 (day 1 of 28 day cycle) up to 18 months
  To document the best combined CR and VGPR rate of first-line treatment with bendamustine and rituximab plus acalabrutinib in patients with WM using response criteria from the Sixth International Workshop on Waldenstrom's Macroglobulinemia9. Response will be documented at cycle 7, 12 and 18 (durable CR).

SECONDARY OUTCOMES:
Overall objective response and partial response | 6 and 12 months
  using criteria from 6th international workshop on WM
Documentation of minimal residual disease (MRD) rate | through study completion, an average of 18 months cycle 7, 12 and 18 (each cycle is 28 days)
  MRD will be assessed at three on treatment timepoints (before start of cycles 7, 12, 18) as well as extended follow-up vistis. MRD will be measured from two body compartments-peripheral blood and bone marrow. MRD will be recorded and will be reported based on the limit of detection of the assay (to be determined). Results will be pooled and rates of MRD negativity for the assay will be recorded at each time point for the pooled patients and for each of the two body compartments that are being assessed.
Documentation of overall survival | Up to 6 years post first dose
  OS will be determined using the time from first day of study treatment to death for each patients. Results for each patient will be pooled to derive an overall survival rate.
Documentation of progression free survival | Up to 6 years post first dose
  PFS will be defined as the time from first dose of study treatment to the first objective documentation of progressive disease (PD), the start of an alternative anticancer therapy, or death from any cause during study. Results for each patient will be pooled to derive an overall progressive free survival rate. Participants not meeting criteria for PD will be followed by telephone every 6 months for up to six years from the time of first dose.
Toxicities graded according to the NCI Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE, v5.0)] | Up to 30 days following last dose
  A descriptive analysis of safety will be performed with descriptions of frequency and grade of the adverse events including adverse events of special interest such as hypertension, cardiac arrhythmias and bleeding events. The common toxicities described in the NCK common terminology criteriae for adverse events (NC CTAE v5.0) will be documented and grade in each patient at each visit throughout the trial. Rates and severity of all of these toxicity will be collected and reported.
Duration of Response | Up to 6 years post first dose
  Defined as the length of time a participant is identified as CR or VGPR until they progress. Different from PFS
Time to Next Treatment | Up to 6 year post first dose
  Defined as the amount of time from the start of trial until the patient requires a new form of treatment to treat their WM

CONTACTS AND LOCATIONS:
Overall Officials: Neil L Berinstein, MD, Principal Investigator — Sunnybrook Research Institute
Locations (9):
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre - Juravinksi, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHU de Quebec - University Laval, Laval, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Aggregate data may be shared